CLINICAL TRIAL: NCT01084096
Title: Trial of the Use of Antenatal Corticosteroids in Developing Countries
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: RTI International (Other); Tulane University School of Medicine (Other); Institute for Clinical Effectiveness and Health Policy (Other); University of Alabama at Birmingham (Other); University Teaching Hospital, Lusaka, Zambia (Other); University of Colorado, Denver (Other); Universidad Francisco Marroquín (Other); Jawaharlal Nehru Medical College (Other); Christiana Care Health Services (Other); Aga Khan University (Other); Columbia University (Other); Indiana University (Other); Moi Univeristy (Other); Lata Medical Research Foundation, Nagpur (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN ACT Study
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Preterm Birth
Keywords: Antenatal Corticosteroids, Preterm Birth, Diffusion
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Eligible women at high risk for preterm birth will be identified and four 6 mg doses of dexamethasone will be administered before delivery.
  Interventions: Behavioral: Increasing use of Antenatal Corticosteroids (ACS)
- Control (No Intervention): Control arm will not receive a specific intervention for comparison.

INTERVENTIONS:
Behavioral: Increasing use of Antenatal Corticosteroids (ACS) — Intervention clusters:
  * Increasing administration of ACS to pregnant women at high risk of preterm birth (HRPB) by providing health providers with kits containing dexamethasone, syringes, and instructions. Eligible women receive four injections of 6 mg dexamethasone from the kit or regimen of choice at the site.
  * Improving identification of women at HRPB by diffusing recommendations for ACS use to health care providers, training health care providers to identify signs of preterm labor and eligibility criteria for ACS use, providing reminders to healthcare providers on the use of the kits, and using a color-coded tape to measure uterine height to estimate gestational age in women at HRPB with unknown gestational age.
  Control clusters: no specific intervention for comparison. Both intervention and control clusters: Birth attendants trained in essential newborn care of LBW infants and instructed to teach mothers how to provide care to premature infants.
  Other Names: Four 6 mg doses of dexamethasone
  Arms: Intervention

SUMMARY:
Multi-country two-arm, parallel cluster randomized controlled trial to reduce neonatal mortality through increasing the rate of antenatal corticosteroid administration to eligible women.

DETAILED DESCRIPTION:
One of the United Nations Millennium Summit goals is to reduce the deaths of children <5 years by two-thirds for 2015 (UN, 2000). Given that 38% of all under-five deaths worldwide occur in the first four weeks of life, the goal seems unattainable unless a significant fraction of the neonatal deaths are prevented (Darmstadt et al., 2005). Thus, the provision of health care during the perinatal period in developing countries is a top priority. Preterm birth is a major cause of neonatal mortality, currently responsible for 28% of the deaths overall. As the contribution of preterm birth to neonatal deaths is well above 50% (MacDorman et al., 2005) in middle and high income countries, it is expected that as low income countries improve their development, the relative importance of this cause will increase. One of the most powerful perinatal interventions to reduce neonatal mortality is the administration of antenatal corticosteroids to pregnant women at high risk of preterm birth.

The primary objective will be to evaluate whether a cluster-level multifaceted intervention, including components to improve the identification of pregnancies at high risk of preterm birth and providing and facilitating the appropriate use of steroids, reduces neonatal mortality at 28 days of life in preterm newborns, compared with the standard delivery of care in selected populations of six African, Asian, and Latin American countries.

ELIGIBILITY:
This is an intent-to-treat design and thus all pregnancy outcomes of women who deliver in the study clusters and provide consent will be collected. Cluster-level inclusion criteria include

* At least 250 deliveries per year.
* Birth attendants within the health cluster will be consented to participate

Participant-level inclusion criteria include all pregnant women living in and delivering in the study cluster who:

* Are between 24 and 36 weeks GA;
* Present with signs of preterm labor, amniotic fluid leakage, hemorrhage, or hypertension;
* Provide consent for injection or present to a facility where it is standard of care.

Exclusion Criteria:

* There will not be any specific exclusion criteria for clusters or participants.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 103117 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Althabe, M.D., Principal Investigator — Institute for Clinical Effectiveness and Health Policy (IECS), Buenos Aires, Argentina
Locations (7):
- Institute for Clinical Effectiveness and Health Policy (IECS), Buenos Aires, Argentina
- Universidad Francisco Marroquin Facultad de Medicina, Guatemala City, Guatemala
- India (2):
  - JN Medical College, Belagavi
  - Lata Medical Research Foundation, Nagpur
- Moi University School of Medicine, Eldoret, Kenya
- Aga Khan University, Karachi, Pakistan
- University of Zambia, Lusaka, Zambia

REFERENCES:
- [Derived] McGoldrick E, Stewart F, Parker R, Dalziel SR. Antenatal corticosteroids for accelerating fetal lung maturation for women at risk of preterm birth. Cochrane Database Syst Rev. 2020 Dec 25;12(12):CD004454. doi: 10.1002/14651858.CD004454.pub4. PMID 33368142
- [Derived] Rohwer AC, Oladapo OT, Hofmeyr GJ. Strategies for optimising antenatal corticosteroid administration for women with anticipated preterm birth. Cochrane Database Syst Rev. 2020 May 26;5(5):CD013633. doi: 10.1002/14651858.CD013633. PMID 32452555
- [Derived] Patel A, Prakash AA, Pusdekar YV, Kulkarni H, Hibberd P. Detection and risk stratification of women at high risk of preterm birth in rural communities near Nagpur, India. BMC Pregnancy Childbirth. 2017 Sep 19;17(1):311. doi: 10.1186/s12884-017-1504-4. PMID 28927395
- [Derived] Goldenberg RL, Thorsten VR, Althabe F, Saleem S, Garces A, Carlo WA, Pasha O, Chomba E, Goudar S, Esamai F, Krebs NF, Derman RJ, Liechty EA, Patel A, Hibberd PL, Buekens PM, Koso-Thomas M, Miodovnik M, Jobe AH, Wallace DD, Belizan JM, McClure EM. The global network antenatal corticosteroids trial: impact on stillbirth. Reprod Health. 2016 Jun 2;13(1):68. doi: 10.1186/s12978-016-0174-4. PMID 27255082
- [Derived] Berrueta M, Hemingway-Foday J, Thorsten VR, Goldenberg RL, Carlo WA, Garces A, Patel A, Saleem S, Pasha O, Chomba E, Hibberd PL, Krebs NF, Goudar S, Derman RJ, Esamai F, Liechty EA, Moore JL, McClure EM, Koso-Thomas M, Buekens PM, Belizan JM, Althabe F. Use of antenatal corticosteroids at health facilities and communities in low-and-middle income countries. Reprod Health. 2016 May 27;13(1):66. doi: 10.1186/s12978-016-0176-2. PMID 27228986
- [Derived] Klein K, McClure EM, Colaci D, Thorsten V, Hibberd PL, Esamai F, Garces A, Patel A, Saleem S, Pasha O, Chomba E, Carlo WA, Krebs NF, Goudar S, Derman RJ, Liechty EA, Koso-Thomas M, Buekens PM, Belizan JM, Goldenberg RL, Althabe F. The Antenatal Corticosteroids Trial (ACT): a secondary analysis to explore site differences in a multi-country trial. Reprod Health. 2016 May 24;13(1):64. doi: 10.1186/s12978-016-0179-z. PMID 27221319
- [Derived] Garces A, McClure EM, Figueroa L, Pineda S, Hambidge KM, Krebs NF, Thorsten VR, Wallace DD, Althabe F, Goldenberg RL. A multi-faceted intervention including antenatal corticosteroids to reduce neonatal mortality associated with preterm birth: a case study from the Guatemalan Western Highlands. Reprod Health. 2016 May 24;13(1):63. doi: 10.1186/s12978-016-0178-0. PMID 27221237
- [Derived] Althabe F, Belizan JM, McClure EM, Hemingway-Foday J, Berrueta M, Mazzoni A, Ciganda A, Goudar SS, Kodkany BS, Mahantshetti NS, Dhaded SM, Katageri GM, Metgud MC, Joshi AM, Bellad MB, Honnungar NV, Derman RJ, Saleem S, Pasha O, Ali S, Hasnain F, Goldenberg RL, Esamai F, Nyongesa P, Ayunga S, Liechty EA, Garces AL, Figueroa L, Hambidge KM, Krebs NF, Patel A, Bhandarkar A, Waikar M, Hibberd PL, Chomba E, Carlo WA, Mwiche A, Chiwila M, Manasyan A, Pineda S, Meleth S, Thorsten V, Stolka K, Wallace DD, Koso-Thomas M, Jobe AH, Buekens PM. A population-based, multifaceted strategy to implement antenatal corticosteroid treatment versus standard care for the reduction of neonatal mortality due to preterm birth in low-income and middle-income countries: the ACT cluster-randomised trial. Lancet. 2015 Feb 14;385(9968):629-639. doi: 10.1016/S0140-6736(14)61651-2. Epub 2014 Oct 15. PMID 25458726
- [Derived] Althabe F, Belizan JM, Mazzoni A, Berrueta M, Hemingway-Foday J, Koso-Thomas M, McClure E, Chomba E, Garces A, Goudar S, Kodkany B, Saleem S, Pasha O, Patel A, Esamai F, Carlo WA, Krebs NF, Derman RJ, Goldenberg RL, Hibberd P, Liechty EA, Wright LL, Bergel EF, Jobe AH, Buekens P. Antenatal corticosteroids trial in preterm births to increase neonatal survival in developing countries: study protocol. Reprod Health. 2012 Sep 19;9:22. doi: 10.1186/1742-4755-9-22. PMID 22992312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18m, 2-arm, parallel, cluster-randomized trial in 7 Global Network sites from Oct 2011-Mar 2014. Health providers in intervention clusters identified women at high risk of preterm birth for antenatal corticosteroids. Overall, 349 and 360 health facilities served intervention and control clusters, respectively; most (260 in each group) were clinics.
Pre-assignment Details: The treatment group for each cluster (and thus all women residing in the cluster) was randomly assigned pretrial (1:1) using a stratified procedure to account for pretrial characteristics. 102 clusters were randomly assigned (51 control:51 intervention). One control cluster withdrew because of unrelated safety concerns prior to study start.
Units Other Than Participants: Geographic Cluster
Groups:
- Intervention Group: Women and their babies residing in geographic clusters assigned to the intervention group. If the woman was identified as high-risk for preterm birth from 24 - 36 weeks' gestational age by the intervention she received one course of four doses of 6 mg of dexamethasone every 12 hours. If identified outside the intervention, she received standard of care.
- Control Group: Women and their babies residing in geographic clusters assigned to the control group. If the woman was identified as high-risk for preterm birth, she received standard of care.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started (Women enrolled in the Global Network Maternal Newborn Health Registry during the ACT trial period.) | 49744; 51 Geographic Cluster | 53373; 51 Geographic Cluster
Completed (Delivery and outcome data available from the GN MNHR.) | 48219; 51 Geographic Cluster | 51523; 50 Geographic Cluster
Not Completed | 1525; 0 Geographic Cluster | 1850; 1 Geographic Cluster
Not completed — Lost to Follow-up | 1501 | 1833
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Woman had a miscarriage | 21 | 17

BASELINE CHARACTERISTICS:
Population: Women enrolled in the Global Network Maternal Newborn Health Registry (MNHR) during the Antenatal Corticosteroid Trial period with delivery and outcome data available from MNHR.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 48,219 | 51,523 | 99742
Age, Customized [Count of Participants; unit: Participants]
  <20 | 5,412 | 6,622 | 12034
  20-35 | 41,003 | 42,938 | 83941
  >35 | 1,741 | 1,895 | 3636
  Missing | 63 | 68 | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48,219 | 51,523 | 99742
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 2,115 | 2,292 | 4407
  Pakistan | 7,714 | 8,202 | 15916
  Guatemala | 5,813 | 3,960 | 9773
  Zambia | 4,279 | 5,739 | 10018
  Kenya | 5,900 | 7,103 | 13003
  India | 22,398 | 24,227 | 46625
Education [Count of Participants; unit: Participants]
  No formal schooling | 11,005 | 11,258 | 22263
  Primary | 17,686 | 19,515 | 37201
  Secondary | 15,528 | 16,170 | 31698
  University | 3,757 | 4,313 | 8070
  Missing | 243 | 267 | 510
Parity [Count of Participants; unit: Participants]
  0 | 16,366 | 17,901 | 34267
  1 | 13,961 | 14,599 | 28560
  2 | 17,570 | 18,934 | 36504
  Missing | 322 | 89 | 411

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Mortality Rate at 28 Days in <5th Percentile Birth Weight Infants (as a Proxy Measure for Prematurity)
Description: Neonatal deaths before 28 days per 1,000 live births among <5th %tile birth weight infants. The <5th %tile birth weight group was a proxy for preterm. Site-specific cutoffs from pretrial data were 2,450g-Argentina, 2,400g-Zambia, 2,267g-Guatemala, 2,000g-Belgaum, India, 2,150g-Pakistan, 2,000g-Nagpur, India, and 2,500g-Kenya. Infants were classified as <5th %tile on the basis of measured birth weights. Estimated weights by clinical assessment were used when measured weights were unavailable; those missing weights were classified as <5th %tile (since based on historical data, most of the missing data were for preterm infants). We used birth weight rather than gestational age (GA) for the primary analysis subgroup because many women in the registry had missing or uncertain GA, ultrasound was often unavailable, and the intervention was designed to improve estimation of GA, which could potentially bias GA-based analyses. All live births, including multiple births, are included.
Time Frame: Birth to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 2,520 | 2,258
Participants | 566 | 524
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority — Trial powered to detect a 30% reduction in 28-d NM among <5th %tile for birth weight infants. We used an intention-to-treat approach, with a model-based adaptation of the permutation test. We fitted an individual-level linear model with 28-d NM by site and randomization strata, nested within site, and computed the residual for each individual and mean cluster-level residuals. Next, we used an ANOVA model to test for trt differences between mean residuals for intervention and control clusters; p = 0.65, t-test, 2 sided; Cluster-level with 62 degrees of freedom [101 clusters-37 strata-2 treatment groups]; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.87 to 1.06] — Calculated from generalized linear models accounting for the cluster-level variance and adjusted for randomization strata. Each stratum corresponds to 2-4 clusters within the site with equal distribution to treatment and control arms

2. Secondary Outcome: Use of Antenatal Corticosteroids in Women at Risk of Preterm Birth in All the Study Clusters
Description: Antenatal corticosteroids provided antepartum assessed in women with a less-than-5th-percentile for birth weight infants. Site-specific cut offs were determined from pretrial data.
Time Frame: 48 hours after identification of risk for preterm birth
Population: Among women with a less-than-5th-percentile for birth weight infant and with data on administration of antenatal corticosteroid data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 2,327 | 2,062
Participants | 1,052 | 215
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; The trial was powered to detect a 30% reduction in 28-day neonatal mortality among infants born at less than the 5th percentile of birth weight, based on previous research and an expected increase from 10% to 50% in the use of antenatal corticosteroids among women at risk of preterm birth in the intervention group; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; P-values were calculated from Cochran-Mantel-Haenszel test controlling for randomization strata; Risk Difference (RD) = 0.3546, 95% CI 2-sided [0.3299 to 0.3792] — Risk difference represents risk in the intervention clusters minus the risk in the control clusters

3. Secondary Outcome: Suspected Maternal Infection
Description: Maternal safety was assessed through the frequency of suspected maternal infection, a composite of process outcomes including receipt of antibiotics plus hospital admission or referral, and receipt of intravenous fluids, surgery, or other treatment related to infection. The definition also included evidence of antepartum or post-partum infection for mothers with infants with a birthweight less than 2500 g. Additionally, use of antenatal corticosteroids, neonatal and perinatal mortality, and suspected maternal infection were measured for all births, irrespective of birthweight.
Time Frame: Pregnancy through 6 weeks postpartum
Population: Women with infection data available from all data sources
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 48,214 | 51,523
Participants | 1,207 | 867
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other — Descriptive analysis; p < 0.0001, Cochran-Mantel-Haenszel — P-values were calculated from Cochran-Mantel-Haenszel test controlling for randomization strata; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.33 to 1.58]

4. Secondary Outcome: Maternal Mortality Rate
Description: The denominator for maternal deaths through 42 days is pregnancy ending in live birth + all maternal deaths. Maternal mortality includes all maternal deaths through 42 days postpartum, irrespective of cause.
Time Frame: Pregnancy through 42 days postpartum
Population: All maternal deaths and pregnancy ending in live birth.
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 46,965 | 50,308
participants | 106 | 97

5. Secondary Outcome: Neonatal Mortality Rate
Description: Number of neonatal deaths before 28 days per 1,000 live births
Time Frame: Birth to 28 days
Population: All live births, including multiples
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 47,394 | 50,743
Participants | 1300 | 1211
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.0127, Generalized linear model with GEE — P-value calculated from a generalized linear model with generalized estimating equations to estimate parameters while controlling for cluster correlations. Model-generated p value was adjusted for randomization strata; Risk Ratio (RR) = 1.12, 95% CI 2-sided [1.02 to 1.22] — Relative risk calculated from a generalized linear model with generalized estimating equations to estimate parameters while controlling for cluster correlations. Model-generated measure of risk was adjusted for randomization strata

6. Secondary Outcome: Stillbirth Mortality Rate
Description: Number of stillbirths per 1,000 births
Time Frame: 20 weeks' gestational age to birth
Population: All births, including multiples.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 48,698 | 52,007
Participants | 1304 | 1264
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other — Descriptive analysis; p = 0.0181, Generalized linear model with GEE — [p-value comment as in outcome 5, analysis 1]; Risk Ratio (RR) = 1.11, 95% CI 2-sided [1.02 to 1.22] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: During the period that the trial was active in a particular cluster, serious adverse events were captured on each woman from the time the woman was enrolled in the MNH registry until 6 weeks after delivery for each pregnant woman enrolled in the MNH registry and her babies.
Description: Total number of serious adverse events is out of all participants (i.e. the number of women plus the number of babies (stillbirths and live births)).
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 2932/48698 | 2774/52007
Other Adverse Events (participants affected / at risk) | 0/48698 | 0/52007
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Intervention Group (N=48698) | Control Group (N=52007)
Maternal death (Pregnancy, puerperium and perinatal conditions) | 50/48219 | 49/51523
Stillbirth/neonatal death (Pregnancy, puerperium and perinatal conditions) | 2604 | 2475
Congenital anomaly (Pregnancy, puerperium and perinatal conditions) | 278 | 250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No